CLINICAL TRIAL: NCT00595205
Title: Post-Authorization Safety Study (PASS) of Post-Marketing Surveillance for Intussusception Following Rotarix™ Introduction Into the Instituto Mexicano Del Seguro Social (IMSS) in Mexico
Brief Title: Intussusception Surveillance After Rotarix Introduction in Mexico
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 104435
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Intussusception (IS); Rotavirus Vaccines
Keywords: vaccination; intussusception; Rotavirus; vaccine
MeSH Terms: conditions — Intussusception

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Group IS: Subjects <1 year of age with definite intussusception cases who had received Rotarix™.
  Interventions: Other: Hospital log review.

INTERVENTIONS:
Other: Hospital log review. — Reviewing of the hospital log to monitor for the occurrence of intussusception.

SUMMARY:
GSK Biologicals' rotavirus vaccine, Rotarix™ has been recommended for universal use targeting infants through the Expanded Program on Immunization (EPI) in Mexico. This protocol describes a Phase IV safety study in Mexico designed to further evaluate the safety profile of Rotarix™ with regard to intussusception (IS). The data generated by this study will be useful for public health officers and policy makers in confirming the safety profile of Rotarix™.

DETAILED DESCRIPTION:
Rationale for amendment 3:

The findings from the first year of the implementation of the active surveillance showed that most Lower Respiratory Tract-Related Post-Neonatal (LRTI) Mortality cases could not be included into the study, because most of the grieving parents refused to participate in the study. The European Medicines Agency Marketing Authorization Holders (EMEA MAH) also generated a substantial amount of additional clinical and post-marketing safety data throughout the world, which clearly indicated the absence of any safety signal when considering the LTRI-related fatalities. Therefore surveillance for LRTI mortality cases was removed from the study design. The number of sites was reduced from approximately 230 to about 60 to 90 in order to reflect the above mentioned change that reduced the need for so many sites. Additionally, passive surveillance for IS cases through the IMSS database was not feasible, due to restrictions of the IMSS internal policies and to the current limitations in the databases linkage and structure abilities.

Lastly, SAEs reporting procedures had to be adjusted according to the Council for International Organizations of Medical Sciences (CIOMS) Working Group V, 2001 publication such that there will be no expedited safety reporting for this study.

Design This is a post marketing ,Phase IV, observational, prospective, self-controlled case series, vaccine safety study including: a) hospital-based surveillance to monitor for the occurrence of IS through active surveillance; b) a self-controlled case series (SCCS) design/analysis to assess the temporal association with Rotarix™ of the IS ascertained through active surveillance.

The aim of the active hospital-based surveillance system is to identify all definite IS cases in children younger than one year of age (children ineligible on day of first birthday) among IMSS members. Surveillance will be conducted in approximately 60 to 90 IMSS health facilities with pediatric surgery service.

Study participation for children fitting the surveillance case definition of IS will include parental/guardian/legal representative interview, as well as a review of medical charts and vaccination records. Additional medical information will be collected through medical record review during hospitalization and after the child has been discharged.

ELIGIBILITY:
Inclusion Criteria:

A child's clinical episode will be defined as an IS case and deemed eligible for the study if he/she meets the following criteria:

* Subject is an IMSS affiliate
* Subject is being treated/has been treated/has been referred for treatment at one of the IMSS hospitals/medical facilities with IS during the study period.
* Male or female child is <one year of age at the time of diagnosis of the IS (child becomes ineligible on the day of their first birthday)
* Subject is diagnosed with definite IS based on the Brighton criteria
* Written informed consent is obtained from the parent/guardian/legal representative of the subject Subjects meeting the above criteria will be eligible for inclusion in this study regardless of whether or not the subject has had a radiographically or surgically confirmed case of IS prior to the current episode.

Exclusion Criteria:

Not applicable

Max Age: 364 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All eligible children < 1 year of age (children ineligible on day of first birthday) who are/have been treated at one of the study hospitals/medical facilities with definite intussusception.
Sampling Method: Non-Probability Sample
Enrollment: 786 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of definite IS episodes within Day 0 to Day 30 following vaccination | 0- 30 days following Rotarix vaccination

SECONDARY OUTCOMES:
Occurrence of definite IS episodes within Day 0 to Day 15 following vaccination | Day 0 to Day 15 post Rotarix vaccination
Yearly occurrence of definite IS episodes (regardless of vaccination status) | Assessed for the interim analysis and after study conclusion

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mexico City, Mexico

REFERENCES:
- [Background] Velázquez FR et al. Postmarketing surveillance to assess risk of intussusception following introduction of the G1P[8] human rotavirus vaccine in Mexico. Abstract presented at the Excellence in Paediatrics (EXPE). London, UK, 2-4 December 2010.